CLINICAL TRIAL: NCT05263596
Title: SARCOPEDIA - Sarcopenia Diagnostics in Aging Medicine
Acronym: SARCOPEDIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-01907
Record Dates: First submitted 2022-02-03; First posted 2022-03-02 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Muscle Weakness; Frailty
MeSH Terms: conditions — Sarcopenia; Muscle Weakness; Frailty | interventions — Absorptiometry, Photon; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Sarcopenia (Control Group) (Other): healthy participants
  Interventions: Diagnostic Test: dual x-ray absorptiometry, body impedance analysis, muscle strength measurements, ultrasound
- Sarcopenia is probable (Other): Low muscle strength (in accordance with the guidlines of "The European Working Group on Sarcopenia in Older People 2" (EWGSOP2))
  Interventions: Diagnostic Test: dual x-ray absorptiometry, body impedance analysis, muscle strength measurements, ultrasound
- Sarcopenia is confirmed (Other): Low muscle strength + low muscle quantity (in accordance with the guidlines of "The European Working Group on Sarcopenia in Older People 2" (EWGSOP2))
  Interventions: Diagnostic Test: dual x-ray absorptiometry, body impedance analysis, muscle strength measurements, ultrasound

INTERVENTIONS:
Diagnostic Test: dual x-ray absorptiometry, body impedance analysis, muscle strength measurements, ultrasound — Results from the routine geriatric assessment:
  * Mini Mental State Exam (MMSE)
  * Clock-drawing test (CDT)
  * Geriatric depression scale (GDS)
  * Functional independence measure (FIM) at admission
  * Timed up and go Test (TUG)
  * Gait speed
  * Hand grip strength (HGS)
  * Nutritional risk screening (NRS)
  Additional measurements:
  * Chair-stand-test
  * Clinical frailty scale (CFS)
  * Calf circumference and mid-arm circumference
  * Body impedance analysis (BIA)
  * US
  * DXA

SUMMARY:
Musculoskeletal aging is one of the major responsibilities and challenges for public health. In particular, sarcopenia correlates with an increased risk of falls and increased morbidity and mortality. With regard to screening for sarcopenia, the guidelines of the European Working Group on Sarcopenia in Older People (EWGSOP2) refer to algorithmic case finding, diagnosis, and quantification of the severity of sarcopenia in clinical. While functional measurements are more difficult to standardize and associated with higher variability, Dual-energy X-ray absorptiometry (DXA) is considered a highly accurate method, even referred to as the "gold standard" to determine muscle mass in the scientific literature. Nevertheless, DXA, which is routinely used, shows inconsistent correlation with functional decline in muscle strength. Another method of muscle quantification is bioelectrical impedance analysis (BIA), a simple, portable instrument that is more readily available and applicable due to its lower cost. However, it tends to overestimate muscle mass and is also more susceptible to a person's hydration status. Because of these difficulties, recent research has focused on the potential of using shear wave elastography. This method indirectly serves to quantify the rapid type II muscle fibers in order to make statements about the muscle quality because an age-related decrease in type II muscle fibers is associated with a more frequent fall frequency.

First, the investigators will define three different categories according to the EWGSOP 2 guidelines based on the muscle strength (grip strength, assessed by pneumatic hand dynamometer) and muscle mass (Appendicular skeletal muscle mass, assessed by BIA): "No Sarcopenia", "Probable Sarcopenia" and "Confirmed Sarcopenia". Within these categories, the Investigators would like to establish a multivariate data analysis of different functional measurements with quantitative imaging results. This exploratory trial design is intended to improve understanding within the three categories and to test proxy measurements of different patients who are ruled out for common routine measurements due to, for example, cognitive impairment or pre-existing rheumatic disease. This is essential to consider the heterogeneity of the aging society proportionally.

DETAILED DESCRIPTION:
Once written informed consent is available, the following data are extracted from the patient's medical records: age and gender, number of medications and number of pre-existing chronic conditions, statin therapy (binary evaluation yes/ no), the laboratory values for CRP, prealbumin, cholinesterase, GFR and CK, and results from geriatric assessment routinely performed by a physiotherapist at admission or a resident physician: Mini Mental State Exam (MMSE), Clock-drawing test (CDT), Geriatric depression scale (GDS), Functional independence measure at admission (FIM) assessed by nurses or physiotherapist. Hand grip strength (HGS), Timed up and go Test (TUG) and Gait speed at admission assessed by physiotherapists; Nutritional risk screening (NRS) assessed by a nutritionist.

To complete baseline data, calf and mid-arm circumference will be measured. Meanwhile, the frailty of the participant is estimated by using the CFS.

For evaluation of muscle mass, body impedance analysis (BIA) is performed in all included patients using a BIVA 101® (Akern, SMT medical GmbH, Würzburg, Germany) within the first 6 days of hospitalization. To conduct this measurement, the patients lie in supine position with extremities stretched, not touching their core and not moving during the measurement. The measurement itself takes only a few seconds. Altogether, the measurements including the preparation phase will be performed within 10 to 15 minutes. As a potential bias, the hydration status of a patient can impair reliability of BIA results. Therefore, all measurements will take part at least 2 hours after the last meal in order to minimize possible fluctuations. If a patient suffers from an altered hydration status at admission (either clinically dehydrated or volume overloaded), the patient will be re-evaluated three days later and BIA measurement will be done if the patient is euvolemic at that time. Concerning those patients receiving continuous enteral feeding, BIA measurement will be performed only if <150 ml/h were delivered in the preceding 2 hours.

For further assessment of muscle mass, non-invasive DXA provides the total body Skeletal Muscle Mass (SMM) and the Appendicular Skeletal Muscle Mass (ASM). For these examinations, the patient cannot stay at her/ his room and will be transferred to an examination room. There an experienced physician will be present if needed for medical assistance before, during or after measurements. The device used for this study is the iDXA densitometer (GE Healthcare, Madison, WI, USA). Here, the study participant moves to an examination couch. The instrument, which is located opposite the examination couch, has an open design and can be viewed from all sides. A narrow scanner runs over the body at a distance of about 20 cm. The examination itself takes about 5 minutes while the patient remains relaxed and calm, breathing normally. In principle, muscle mass is correlated with body size, i.e. persons with a larger body size usually have a larger muscle mass. Therefore, when quantifying muscle mass, the absolute level of SMM or ASM can be adjusted for body size in several ways, namely by using height squared (ASM/height2), weight (ASM/weight), or body mass index (ASM/BMI), all of which are included in the assessment. As a definition of sarcopenia, cut-off points from EWGSOP2 will be used. All precision scans are performed by the same radiologic technologist under the supervision of the project manager.

A subsequent ultrasound examination (Philips PureWave EPIQ 5G, Amsterdam, Netherlands) will be used to detect the elasticity via elastography of two muscles in defined positions. The measurements positions are the Musculus (M.) quadriceps femoris in a supine position on an examination couch and the M. biceps brachii in an elbow flexed position at 90° with the forearm rested on the body. The probe will be placed on top of the skin with a minimal load ensuring no external pressure could affect the measurements. The elastography will be recorded in kilopascals (kPa). The examination, which takes about 5 minutes is also completely painless, and will be performed by the project leader.

The CST is then performed under the supervision and guidance of the examining physician. This clinical test is also used to assess mobility and is estimated to take approximately 3 minutes.

ELIGIBILITY:
Inclusion Criteria:

The investigators aim to include patients ≥ 65 years old newly admitted for study eligibility at the UAFP.

Exclusion Criteria:

* Lack of informed written consent
* Implanted defibrillation device
* Implanted pacemaker
* Acute sepsis or severe volume overload
* Life expectancy of < 3 months according to treating doctor
* bedridden
* Plasters or bandages that cannot be removed from the feet or hands
* Isolated patients (contact and aerosol)
* Measurement is not possible due to organizational reasons
* Inability to follow the procedures, e.g. due to language problems, psychological disorders

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
No Sarcopenia (healthy participants) - according to the current European Working Group on Sarcopenia in Older People 2 | 12 months
  Normal muscle strength and normal size of muscle masss according to the current European Working Group on Sarcopenia in Older People 2. Grip strength is measured on the dominant hand by a pneumatic hand dynamometer (Martin Vigorimeter) in kPa. Healthy women: ≥ 27 kPa; healthy men: ≥ 45 kPa. Appendicular skeletal muscle mass (ASMM) is measured by the Body Impedance Analysis (BIA 101 Akern, Florence, Italy). Cut-off points for low appendicular skeletal muscle mass index (ASMI), calculated from ASMM/height2, were <7 kg/m2 for men and <5.5 kg/m2 for women
Probable Sarcopenia - according to the current European Working Group on Sarcopenia in Older People 2 | 12 months
  Low muscle strength and normal size of muscle mass according to the current European Working Group on Sarcopenia in Older People 2. Grip strength is measured on the dominant hand by a pneumatic hand dynamometer (Martin Vigorimeter) in kPa. Low muscle strength women: < 27 kPa; low muscle strength men: < 45 kPa. Appendicular skeletal muscle mass (ASMM) is measured by the Body Impedance Analysis (BIA 101 Akern, Florence, Italy). Cut-off points for low appendicular skeletal muscle mass index (ASMI), calculated from ASMM/height2, were <7 kg/m2 for men and <5.5 kg/m2 for women
Confirmed Sarcopenia - according to the current European Working Group on Sarcopenia in Older People 2 | 12 months
  Low muscle strength and low muscle mass according to the current European Working Group on Sarcopenia in Older People 2. Grip strength is measured on the dominant hand by a pneumatic hand dynamometer (Martin Vigorimeter) in kPa. Low muscle strength women: < 27 kPa; low muscle strength men: < 45 kPa. Appendicular skeletal muscle mass (ASMM) is measured by the Body Impedance Analysis (BIA 101 Akern, Florence, Italy). Cut-off points for low appendicular skeletal muscle mass index (ASMI), calculated from ASMM/height2, were <7 kg/m2 for men and <5.5 kg/m2 for women

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M. Fischer, Principal Investigator — Universitäre Altersmedizin Felix Platter
Locations (1):
- Universitäre Altersmedizin Felix Platter, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Van Ancum JM, Scheerman K, Jonkman NH, Smeenk HE, Kruizinga RC, Meskers CGM, Maier AB. Change in muscle strength and muscle mass in older hospitalized patients: A systematic review and meta-analysis. Exp Gerontol. 2017 Jun;92:34-41. doi: 10.1016/j.exger.2017.03.006. Epub 2017 Mar 10. PMID 28286250
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372